CLINICAL TRIAL: NCT00903539
Title: Prospective SecurAcath Subcutaneous Securement Clinical Trial
Brief Title: Prospective SecurAcath Subcutaneous Securement Trial
Acronym: SecurAcath
Status: Completed | Type: Observational
Sponsor: Interrad Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 1180-001
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Central Venous Catheter
Keywords: Peripherally Inserted Central Catheter; Central Venous Catheter; Intravenous Catheter; StatLock; Patients indicated to have an intravenous catheter placed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SecurAcath Securement System — Subcutaneous catheter securement system
  Other Names: PICC securement system

SUMMARY:
To prospectively monitor the safety and performance of the catheter securement device in subjects whose catheter is secured with the Interrad Medical SecureAcath device.

DETAILED DESCRIPTION:
Peripherally inserted central catheters (PICCs) and Central Venous Catheter (CVC) are widely used to deliver fluids directly to the central venous system and can remain in place for as short as a few days to as long as months. One of the highest risks in the use of these catheters is infection, both local and systemic. Currently, these catheters are secured by either sutures or adhesive patches. Sutures can create additional potential entry points for bacteria whereas both sutures and adhesive securement patches hold the catheter hub to the skin resulting in increased difficulty cleaning around the catheter entry site. Furthermore, securing a catheter outside the skin away from the catheter entry point, as with sutures or adhesive securement patches may potentiate pistoning of the catheter which is also believed to possibly increase infection risks. A second risk of intravenous catheter use is dislodgement during normal use and site maintenance. These catheters are often manipulated multiple times a day for blood sampling or injection of fluids. During manipulation, the catheter can be dislodged thus requiring an unplanned replacement of the catheter.

Interrad Medical has developed a means to secure indwelling catheters using a small subcutaneous anchor. With this system, cleaning around the catheter entry site is made easier and can be more thorough. The system is also designed to minimize the risk of catheter dislodgement because once the anchor is deployed, the catheter remains secured. This may simplify dressing changes compared to adhesive devices such as Statlock, which requires the catheter be released from the device and therefore be unsecured during dressing changes.

The objective of this post-market study is to monitor the safety and performance of the SecurAcath when used to secure the catheter to the insertion site via a subcutaneous anchor. The data collected may provide insight for future enhancements to improve the safety and utility of the device. It also provides a means for an early warning of any identified safety issues, and allows physicians to share their experiences thereby improve the quality of care provided to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Requires an intravenous catheter to be placed

Exclusion Criteria:

* Inability to understand the study or a history of non-compliance with medical advice.
* Unwilling or unable to sign Informed Consent Form (ICF).
* Had a previous catheter placed in the same side within the last 3 months.
* Known central venous thrombosis or occlusion or stenosis on the side of the body to be used for the catheter.
* History of upper extremity venous thrombosis on the side of the body to be used for the catheter.
* Known hypercoagulable disorder.
* Diffuse skin inflammatory condition or rashes on the side to be used for the catheter line.
* Peripheral chemotherapy therapy in the same side as that to be used for the catheter line within 3 months.
* Known hypersensitivity to nickel.
* Any infection associated with positive blood cultures that are still present after 48 hours of antibiotic therapy.
* Previous mastectomy or axillary lymph node dissection on the same side as catheter implant.
* Subjects on chronic or recurrent systemic steroid medications for 6 months or longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated to have a central catheter placed at a hospital or private practice clinic are included in the study population.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Device Securement Success: defined as the percent of devices implanted and explanted without malfunction or device related complications attributed to the subcutaneous securement system. | Timeframe is the length of time the patient has the catheter in place. Can vary depending on the indication for the catheter (anywhere from 48 hours post-procedure to 6 months or more).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - North Memorial Hospital - Minneapolis Radiology, Robbinsdale, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - Great Basin Imaging, Carson City, Nevada
  - Albany Medical Center, Albany, New York